CLINICAL TRIAL: NCT00499863
Title: A Phase IIIb, Randomized, Double-Blind, Multi-Center, Parallel-Group, Placebo-Controlled, Dose Optimization Study, Designed to Evaluate the Efficacy and Safety of MTS in Adolescents Aged 13-17 Years With ADHD
Brief Title: Evaluate the Efficacy &Safety of Methylphenidate Transdermal System (MTS) in Adolescents Aged 13-17 Years With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD485-409
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2009-06-11 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate Transdermal System (Experimental): dose optimization of 4 doses of the MTS transdermal patch over the same duration of wear
  Interventions: Drug: methylphenidate transdermal system
- 2 (Placebo Comparator): Daily application of matching MTS Placebo Patch
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methylphenidate transdermal system — dose optimization of 4 doses of the MTS transdermal patch over the same duration of wear
  Other Names: DAYTRANA
  Arms: Methylphenidate Transdermal System
Drug: Placebo — Placebo patch
  Other Names: Sham treatment
  Arms: 2

SUMMARY:
To assess the efficacy and safety of efficacy of MTS compared to placebo

DETAILED DESCRIPTION:
To assess the efficacy and safety of efficacy of MTS compared to placebo, as determined by the change in the clinician completed ADHD Rating Scale - Version 4th Edition (ADHD-RS-IV), in the symptomatic treatment of adolescents (aged 13-17 years) diagnosed with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must meet criteria for a primary diagnosis of ADHD based on a detailed psychiatric evaluation.
2. Subject must have a total score of ≥26 on the ADHD-RS-IV at the Baseline Visit (Visit 2).
3. Subject must have a minimum level of intellectual functioning, as determined by an IQ (based on Kaufman Brief Intelligence Test [KBIT]) score of 80 or above.
4. Subject has blood pressure measurements within the 95th percentile for age, gender, and height at Screening and Baseline.
5. Subject is a male or female aged 13 17 years.
6. Females must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test at Screening and a negative urine pregnancy test at Baseline and agree to use acceptable contraceptives throughout the study period and for 30 days after the last dose of IP.

Exclusion Criteria:

1. Subject has a current, controlled (requiring a restricted medication) or uncontrolled, with significant symptoms such as Post Traumatic Stress Disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder.
2. Subjects who, in the opinion of the Investigator, are acutely at risk for suicidal or violent behavior towards him/herself or others, or a history of a suicide attempt requiring medical intervention.
3. Subject is overweight.
4. Subject has a history of seizures during the last 2 years, a tic disorder, a current diagnosis and/or family history of Tourette's Disorder.
5. Subject has Conduct Disorder.
6. Subject has a positive urine drug or alcohol result at Screening (with the exception of subject's current stimulant therapy, if any).
7. Subject has a history of alcohol or other substance abuse or dependence.
8. Subject has taken an investigational drug within 30 days prior to screening.
9. Subject has any abnormal thyroid function.
10. Subject has any clinically significant laboratory abnormalities.
11. Subject has severe allergic rhinitis, disability, or other condition that might confound the results of safety assessments administered in the study or that might increase risk to the subject. Mild, stable asthma is not exclusionary.
12. The female subject is pregnant or lactating.
13. Subject has any skin disease, or history of any chronic skin disease, skin cancer, skin manifestations of allergic disease, or other dermatologic conditions which would interfere with trial assessments or compromise subject safety (e.g. dermatitis, eczema or psoriasis).
14. Subject has sensitive-skin syndrome (definition: subjects who often develop nonspecific skin irritancy reactions to bland materials) or has sensitivities to the ingredients in soaps, lotions, cosmetics or adhesives.
15. Subject has clinical signs and symptoms of skin irritation (i.e., pruritus, burning, erythema) or scars or tattoos.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Finding, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (32):
- United States (32):
  - Melmed Center, Scottsdale, Arizona
  - Bay Area Research Institute, Lafayette, California
  - Elite Clinical Trials Inc., Wildomar, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Miami Research Associates, South Miami, Florida
  - Northwest Behavioral Research Ctr, Roswell, Georgia
  - Mountain West Clinical Trials, LLC, Eagle, Idaho
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Shire Clinical Research Site, Lexington, Kentucky
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Clinical Neurophysiology Services, PC, Troy, Michigan
  - CRI Worldwide, Clementon, New Jersey
  - Triangle Neuropsychiatry, Durham, North Carolina
  - Dakota Clinic/Innovis health, Fargo, North Dakota
  - Odyssey Research, Minot, North Dakota
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oregon Center for Clinical Investigations, Inc., Eugene, Oregon
  - OCCI, Inc, Portland, Oregon
  - Shire Clinical Research Site, Media, Pennsylvania
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - CNS Healthcare, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Claghorn-Lesem Research, Ltd., Bellaire, Texas
  - Westex Clinical Investigations, Lubbock, Texas
  - Cerebral Research, LLC, San Antonio, Texas
  - Vermont Clinical Study Center, Burlington, Vermont
  - NeuroScience, Inc., Herndon, Virginia
  - Adolescent Health Center, Midlothian, Virginia
  - Northwest Clinical Research Center, Friday Harbor, Washington
  - Eastside Therapeutic Resource, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Findling RL, Turnbow J, Burnside J, Melmed R, Civil R, Li Y. A randomized, double-blind, multicenter, parallel-group, placebo-controlled, dose-optimization study of the methylphenidate transdermal system for the treatment of ADHD in adolescents. CNS Spectr. 2010 Jul;15(7):419-30. doi: 10.1017/s1092852900000353. PMID 20625364

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 217 subjects were enrolled and randomized. The study included a screening/washout period, a 5 week dose optimization period, a 2 week maintenance period, and a follow-up period.
Groups:
- Methylphenidate Transdermal System: Methylphenidate Transdermal System Patch
- Placebo (PTS): Placebo Transdermal System
Period: Overall Study
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Started | 145 | 72
Completed | 95 | 29
Not Completed | 50 | 43
Not completed — Lack of Efficacy | 21 | 27
Not completed — Protocol Violation | 12 | 7
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Adverse Event | 8 | 2
Not completed — Sponsor decision | 2 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS) | Total
Number analyzed (Participants) | 145 | 72 | 217
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 145 | 72 | 217
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.25) | 14.6 (1.42) | 14.6 (1.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 19 | 55
  Male | 109 | 53 | 162
Region of Enrollment [Number; unit: participants]
  United States | 145 | 72 | 217

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Attention Deficit Hyperactivity Disorder Rating Scale-fourth Edition (ADHD-RS-IV) Total Score at Endpoint
Description: The Attention Deficit Hyperactivity Disorder Rating Scale-fourth edition (ADHD-RS-IV) consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: baseline and endpoint (up to 7 weeks)
Population: Intent-to-treat (ITT) which included all randomized subjects who received at least one dose of MTS or PTS, and had one Baseline and at least one post-Baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 143 | 72
scores on a scale | -18.8 (1.01) | -8.8 (1.42)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System vs Placebo (PTS); The null hypothesis was that there is no difference between MTS and placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Change From Baseline in the Conner's Parent Rating Scale-Revised (CPRS-R) Total Score at Endpoint
Description: The Conner's Parent rating Scale-revised short version (CPRS-R) consists of 27 questions graded on a scale from 0 (not true at all) to 3 (very much true).
Time Frame: Baseline and endpoint (up to 7 weeks)
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 143 | 72
scores on a scale | -20.9 (1.45) | -7.5 (2.08)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System vs Placebo (PTS); Test type: Superiority or Other; p < 0.001, ANCOVA

3. Secondary Outcome: Improvement in Clinical Global Impressions-Improvement (CGI-I) Score
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement includes a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: up to 7 weeks
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 143 | 72
Participants | 93 | 22
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System vs Placebo (PTS); Test type: Superiority or Other; p < 0.001, Chi-squared

4. Secondary Outcome: Improvement in Parent Global Assessment (PGA) Score
Description: Parent Global Assessment (PGA) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement includes a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: up to 7 weeks
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 143 | 72
Participants | 76 | 15
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System vs Placebo (PTS); Test type: Superiority or Other; p < 0.001, Chi-squared

5. Secondary Outcome: Change From Baseline in Youth Quality of Life-research Version (YQOL-R) Total Score at Endpoint
Description: The Youth Quality of Life Instrument-research version (YQOL-R) is a validated 56-item generic instrument for comparing quality of life of adolescents across condition groups that scores each question on a scale from 0 (never) to 4 (very often).
Time Frame: Baseline and endpoint (up to 7 weeks)
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 143 | 72
scores on a scale | 3.3 (1.06) | 1.3 (1.55)
Statistical Analysis 1: Comparison: Methylphenidate Transdermal System vs Placebo (PTS); Test type: Superiority or Other; p = 0.288, ANCOVA

6. Other Pre Specified Outcome: Post Sleep Questionnaire (PSQ) Quality of Sleep
Description: Post Sleep Questionnaire (PSQ) overall rating of quality of sleep. There are 5 rating responses ranging from very poor to very good. No numbers are associated with the rating responses.
Time Frame: up to 7 weeks
Population: Safety population (Note: not everyone in the safety population completed a sleep questionnaire)
Measure: Number; unit: Participants
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 145 | 72
Participants
  Very poor | 2 | 2
  Poor | 14 | 7
  Average | 27 | 13
  Good | 47 | 18
  Very good | 31 | 18

7. Secondary Outcome: Dermal Response Scale (DRS) Scores
Description: Mean dermal reaction scores were graded on a scale ranging from 0 (no irritation) to 7 (strong reaction) for observed findings of erythema, edema, papules, and vesicles.
Time Frame: up to 7 weeks
Population: Safety population which included all randomized subjects that received at least one dose of MTS or PTS.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 145 | 72
scores on a scale | 0.6 (0.75) | 0.2 (0.66)

8. Secondary Outcome: Change From Baseline in Electrocardiogram Results(QTcF Interval) at Endpoint
Description: QTcF is the QT interval using Fridericia's correction formula. QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate(e.g., the faster the heart rate, the shorter the QT interval). The QT interval has to be corrected in order to aid interpretation.
Time Frame: Baseline and endpoint (up to 7 weeks)
Population: Safety population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 145 | 72
msec | -1.3 (16.70) | -0.8 (13.35)

9. Secondary Outcome: Change From Baseline in Pulse Rate at Endpoint
Time Frame: Baseline and endpoint (up to 7 weeks)
Population: Safety population
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 145 | 72
bpm | 6.5 (11.65) | -1.4 (9.84)

10. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Endpoint
Time Frame: Baseline and endpoint (up to 7 weeks)
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 145 | 72
mmHg | 2.0 (9.44) | -0.4 (11.04)

11. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Endpoint
Time Frame: Baseline and endpoint (up to 7 weeks)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 143 | 72
mmHg | 1.9 (8.00) | 1.1 (8.55)

12. Secondary Outcome: Change From Baseline in Weight at Endpoint
Time Frame: Baseline and endpoint (up to 7 weeks)
Population: Safety population
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Number analyzed (Participants) | 145 | 72
lbs | -1.9 (3.87) | 1.77 (4.38)

ADVERSE EVENTS:
Arm/Group | Methylphenidate Transdermal System | Placebo (PTS)
Serious Adverse Events (participants affected / at risk) | 1/145 | 1/72
Other Adverse Events (participants affected / at risk) | 125/145 | 28/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate Transdermal System (N=145) | Placebo (PTS) (N=72)
syncope (Nervous system disorders) | 1 (2) | 0 (0)
negativism (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate Transdermal System (N=145) | Placebo (PTS) (N=72)
Nausea (Gastrointestinal disorders) | 14 (14) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 7 (7)
Weight decreased (Investigations) | 8 (9) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 37 (41) | 1 (1)
Dizziness (Nervous system disorders) | 8 (8) | 1 (1)
Headache (Nervous system disorders) | 18 (20) | 9 (9)
Insomnia (Psychiatric disorders) | 9 (11) | 2 (2)
Irritability (Psychiatric disorders) | 16 (16) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.